CLINICAL TRIAL: NCT00810888
Title: The Spot Sign for Predicting and Treating Intracerebral Hemorrhage Growth Study
Brief Title: The Spot Sign for Predicting and Treating ICH Growth Study
Acronym: STOP-IT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Matthew Flaherty, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P50NS044283_STOP_IT; 2P50NS044283 (NIH)
Record Dates: First submitted 2008-12-15; First posted 2008-12-18 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-02

CONDITIONS: Intracerebral Hemorrhage
Keywords: intracerebral hemorrhage; ICH; computed tomography angiography; CTA; recombinant activated factor seven; rFVIIa; NovoSeven; recombinant activated factor VII
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1-Recombinant activated factor VII (Active Comparator): Participants with ICH determined by CTA to be high risk for hemorrhage growth ("spot sign" positive for contrast leakage within the brain hematoma) randomized to receive rFVIIa at 80 mcg/kg (max dose 21.3 mL).
  Interventions: Drug: recombinant activated factor VII
- Group 2 - Placebo (Placebo Comparator): Participants with ICH determined by CTA to be high risk for hemorrhage growth ("spot sign" positive for contrast leakage within the brain hematoma) will be randomized to receive placebo.
  Interventions: Drug: placebo
- Group 3 - Observation Only Arm (No Intervention): Participants with ICHdetermined by CTA not to be at high risk for hemorrhage growth (CTA "spot sign" negative) enrolled into a prospective observational group.

INTERVENTIONS:
Drug: recombinant activated factor VII — Participants will receive rFVIIa at 80 mcg/kg (maximum dose volume 21.3 mL, equivalent to maximum weight of 160 kg).
  Arms: Group 1-Recombinant activated factor VII
Drug: placebo — An inactive substance (maximum dose volume 21.3 mL, equivalent to maximum weight of 160 kg)
  Arms: Group 2 - Placebo

SUMMARY:
The purpose of this study is to determine if computed tomography angiography can predict which individuals with intracerebral hemorrhage will experience significant growth in the size of the hemorrhage. For individuals who are at high risk for hemorrhage growth, the study will compare the drug recombinant activated factor VII (rFVIIa) to placebo to determine the effect of rFVIIa on intracerebral hemorrhage growth.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH)-breakage of a blood vessel with bleeding in the brain-is a devastating form of stroke with a 40-50 percent fatality rate and no proven treatment. Because the majority of deaths from ICH occur within several days of the stroke, interventions for improving outcomes must occur early in the treatment course. Among the potentially modifiable determinants of ICH outcome, hematoma growth is a particularly attractive target for intervention and a major focus of this trial.

The purpose of this study is to determine if an imaging test called computed tomography angiography (CTA) can predict which individuals with ICH will experience significant growth in the size of the hemorrhage. Growth of the hemorrhage can cause additional injury and may worsen the outcome. For individuals who are at high risk for hemorrhage growth based on CTA results (i.e., a positive CTA "spot sign," evidence of contrast leakage within the hemorrhage), the study will compare the effects of a drug called recombinant activated factor VII (NovoSeven®) or rFVIIa with a placebo to determine which is better for reducing ICH growth.

The primary goals of this trial are (1) to determine the sensitivity and specificity of the CTA spot sign for predicting hematoma growth; (2) to determine the feasibility of using CTA to identify individuals with ICH who are at high risk of hematoma growth and to select study participants for randomization to treatment with rFVIIa or placebo; and (3) to determine the rate of hematoma growth among spot-positive individuals at 24 hours-comparing individuals treated with rFVIIa to those treated with placebo.

Approximately 184 persons with ICH will be enrolled in one of two study groups at 12 clinical sites across the United States and Canada. Participants with ICH who are determined by CTA to be at high risk for hemorrhage growth (CTA "spot sign" positive) will be randomized to receive either the active study medication, rFVIIa, at 80 mcg/kg, or to receive a placebo (an inactive substance). Participants with ICH who are determined by CTA not to be at high risk for hemorrhage growth (determined to be CTA "spot sign" negative) will be enrolled into a prospective observational group.

Duration of the study for participants is approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Acute, spontaneous ICH (including bleeding in cerebellum) diagnosed by non-enhanced CT scan within five hours of symptom onset. (Time of onset is defined as the last time the patient was witnessed to be at baseline (i.e., subjects who have stroke symptoms upon awakening will be considered to have their onset at beginning of sleep)
* Age >/= 18 years through 80 years (candidates must have had their 18th birthday, but not had their 81st birthday)
* For spot positive patients, dosing of study drug within 90 minutes of enrolling CT scan

Exclusion Criteria:

* Time of symptom onset of ICH is unknown or more than five hours prior to baseline CT scan,
* ICH secondary to known or suspected trauma, aneurysm, vascular malformation, hemorrhagic conversion of ischemic stroke, venous sinus thrombosis, thrombolytic treatment of any condition (e.g., myocardial infarction, cerebral infarction, etc.), central nervous system (CNS) tumor or CNS infection
* Brainstem location of hemorrhage (patients with cerebellar hemorrhage may be enrolled)
* Serum creatinine > 1.4 mg/dl (123 μmol/L). Sites that currently perform CTA as standard of care for ICH will follow their standard procedures regarding renal insufficiency.
* Known allergy to iodinated contrast media
* Intravenous or intra-arterial administration of iodinated contrast media within the previous 24 hours of baseline CT scan
* Known hereditary (e.g., hemophilia) or acquired hemorrhagic diathesis, coagulation factor deficiency, or anticoagulant therapy with international normalized ration (INR) > 1.2
* Known or suspected thrombocytopenia (unless current platelet count documented above 50,000 / μl)
* Unfractionated heparin use with abnormal partial thromboplastin time (PTT)
* Low-molecular weight heparin use within the previous 24 hours
* GPIIb/IIIa antagonist use in the previous two weeks
* Direct thrombin inhibitor or factor Xa inhibitor within the previous 48 hours
* Glasgow Coma Scale score < 8 at time of proposed enrollment
* Pre-admission modified Rankin Scale score > 2
* Baseline ICH volume of < 0.5 cc (Hematoma volume will be estimated by local investigators from the baseline CT using the "ABC / 2 method".)
* Baseline ICH volume of > 90 cc
* Planned surgical evacuation of ICH within 24 hours of symptom onset (placement of intraventricular catheter is not a contraindication to study enrollment.)
* Evidence of acute or subacute ischemic stroke on baseline qualifying CT scan
* Clinical history of thromboembolism or ischemic vascular disease, including myocardial infarction, coronary artery bypass surgery, cardiac angina, transient ischemic attack, ischemic stroke, peripheral artery disease (vascular claudication), cerebral bypass surgery, carotid endarterectomy, deep venous thrombosis, pulmonary embolism, or coronary or cerebrovascular angioplasty or stenting. (Clinically silent evidence of old ischemia on EKG (Q waves) or CT scan (silent old infarct) will not be considered reasons for exclusion.)
* Baseline electrocardiogram shows evidence of acute cardiac ischemia (ST elevation in two contiguous leads, new left bundle branch block (LBBB), or ST depression)
* Clinical history suggestive of acute cardiac ischemia (e.g., chest pain)
* Abnormal baseline troponin
* Females of childbearing potential who are known to be pregnant and/or lactating or who have positive pregnancy tests on admission
* Advanced or terminal illness or any other condition the investigator feels would pose a significant hazard to the patient if rFVIIa were administered
* Recent (within 30 days) participation in any investigational drug or device trial or earlier participation in any investigational drug or device trial for which the duration of effect is expected to persist until the time of STOP-IT enrollment
* Planned withdrawal of care or comfort care measures
* Patient known or suspected of not being able to comply with trial protocol (e.g., due to alcoholism, drug dependency or psychological disorder)
* Informed consent cannot be obtained from the patient or legally authorized representative

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L. Flaherty, MD, Principal Investigator — University of Cincinnati; Edward C. Jauch, MD, MS, Principal Investigator — Primary Emergency Medicine Investigator, Medical University of South Carolina
Locations (10):
- United States (8):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California, San Diego, San Diego, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - University of Cincinnati-Clinical Coordinating Center, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Sunnybrook Health Science Center, Toronto, Ontario

REFERENCES:
- [Derived] Gladstone DJ, Aviv RI, Demchuk AM, Hill MD, Thorpe KE, Khoury JC, Sucharew HJ, Al-Ajlan F, Butcher K, Dowlatshahi D, Gubitz G, De Masi S, Hall J, Gregg D, Mamdani M, Shamy M, Swartz RH, Del Campo CM, Cucchiara B, Panagos P, Goldstein JN, Carrozzella J, Jauch EC, Broderick JP, Flaherty ML; SPOTLIGHT and STOP-IT Investigators and Coordinators. Effect of Recombinant Activated Coagulation Factor VII on Hemorrhage Expansion Among Patients With Spot Sign-Positive Acute Intracerebral Hemorrhage: The SPOTLIGHT and STOP-IT Randomized Clinical Trials. JAMA Neurol. 2019 Dec 1;76(12):1493-1501. doi: 10.1001/jamaneurol.2019.2636. PMID 31424491
- See also: trial website — http://www.STOPITSTUDY.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 - Randomized to Study Drug: Participants with ICH who are determined by CTA to be at high risk for hemorrhage growth (or determined to be CTA "spot sign" positive for contrast leakage within the brain hematoma) will be randomized to receive either rFVIIa at 80 mcg/kg (maximum dose volume 21.3 mL, equivalent to maximum weight of 160 kg) or a placebo .
  Recombinant activated factor VII: Participants will receive rFVIIa at 80 mcg/kg (maximum dose volume 21.3 mL, equivalent to maximum weight of 160 kg).
- Group 2 - Randomized to Placebo: Participants with ICH who are determined by CTA to be at high risk for hemorrhage growth (or determined to be CTA "spot sign" positive for contrast leakage within the brain hematoma) will be randomized to receive either rFVIIa at 80 mcg/kg or a placebo (maximum dose volume 21.3 mL, equivalent to maximum weight of 160 kg).
  Placebo: An inactive substance (maximum dose volume 21.3 mL, equivalent to maximum weight of 160 kg)
- Group 3 - Observation Only Arm: Participants with ICH who are determined by CTA not to be at high risk for hemorrhage growth (determined to be CTA "spot sign" negative) will be enrolled into a prospective observational group.
Period: Overall Study
Arm/Group | Group 1 - Randomized to Study Drug | Group 2 - Randomized to Placebo | Group 3 - Observation Only Arm
Started | 10 | 9 | 73
Completed | 10 | 9 | 73
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population consists of 19 subjects diagnosed as "Spot Positive" on CT and were eligible for randomization within the clinical trial portion of the protocol. In addition 73 subjects diagnosed as "Spot Negative" on CT were followed prospectively with no study intervention. All 92 subjects were followed to 90 days post stroke.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Randomized to Study Drug | Group 2 - Randomized to Placebo | Group 3 - Observation Only Arm | Total
Number analyzed (Participants) | 10 | 9 | 73 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (13.1) | 62.4 (12.2) | 60.7 (34.7) | 61.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 29 | 38
  Male | 4 | 6 | 44 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 17 | 23
  White | 9 | 4 | 56 | 69
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 1 | 23 | 27
  United States | 7 | 8 | 50 | 65
Modified Rankin Score (mRS) [Count of Participants; unit: Participants] — Measure of mobility prior to stroke (0=best, 5=worst)
  Participants
    0 | 10 | 6 | 65 | 81
    1 | 0 | 3 | 6 | 9
    2 | 0 | 0 | 2 | 2
Glasgow Coma Score/Scale (GCS) [Median (Inter-Quartile Range); unit: units on a scale] — Scale to measure severity due to coma status (0=worst, 15=best)
  units on a scale | 15 [14 to 15] | 15 [14 to 15] | 15 [14 to 15] | 15 [14 to 15]
National Institute of Health Stroke Scale (NIHSS) Score [Mean (Standard Deviation); unit: units on a scale] — The National Institute of Health Stroke Scale (NIHSS) Score is a scale which measures stroke severity (0=best, 42=worst)
  units on a scale | 14.1 (3.9) | 12.1 (4.9) | 10.3 (6.2) | 10.9 (6.0)
Time from Stroke to Computed Tomography (CT) Scan [Mean (Standard Deviation); unit: minutes] | 158.8 (77.0) | 90.2 (49.9) | 159.8 (81.9) | 152.9 (80.9)
Time from Stroke to Study Drug Administration [Mean (Standard Deviation); unit: minutes] — Population: The Observational group did not receive study drug so the variable "Time from stroke to study drug administration" is not applicable
  minutes
    number analyzed (Participants) | 10 | 9 | 0 | 19
    (all) | 269.9 (68.3) | 181.1 (47.1) |  | 222.5 (70.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Subjects With Life-threatening Thromboembolic Complications
Description: Thromboembolic complications are defined as development of (1) acute myocardial ischemia; or (2) acute cerebral ischemia; or (3) acute pulmonary embolism
Time Frame: through day 4 after completion of study drug administration
Population: The analysis population consists of 19 subjects diagnosed as "Spot Positive" on CT who were eligible for randomization within the clinical trial portion of the protocol, as well as 73 subjects diagnosed as "Spot Negative" on CT who were followed prospectively with no study intervention. Statistical comparison involves only Group1 and Group 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Randomized to Study Drug | Group 2 - Randomized to Placebo | Group 3 - Observation Only Arm
Number analyzed (Participants) | 10 | 9 | 73
Participants | 1 | 0 | 0
Statistical Analysis 1: Comparison: Group 1 - Randomized to Study Drug vs Group 2 - Randomized to Placebo; Fisher's exact test; Test type: Superiority; p = 1.00, Fisher Exact — not adjusted for multiple comparisons as a prior hypothesis critical value <0.05

2. Primary Outcome: Number of Subjects With Hematoma Growth Among Spot Sign Positive Subjects at 24 Hours.
Description: Comparison of only the subjects with a positive spot sign with respect to a categorical measure of hematoma growth from baseline to 24 hours. the outcome of interest is the percent of subjects with hematoma growth > 33% or > 6 cc increase in volume, from baseline to 24 hours.
Time Frame: From baseline to 24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Randomized to Study Drug | Group 2 - Randomized to Placebo | Group 3 - Observation Only Arm
Number analyzed (Participants) | 10 | 9 | 73
Participants | 4 | 5 | 8
Statistical Analysis 1: Comparison: Group 1 - Randomized to Study Drug vs Group 2 - Randomized to Placebo; Only the randomized subjects will be compared; Test type: Superiority; p = 0.66, Fisher Exact

3. Primary Outcome: The Sensitivity of the Spot Sign for Predicting Hematoma Growth
Description: The outcome measure is hematoma growth. Groups 2 and 3 only will be compared as Group 1 had administration of study drug which was hypothesized to reduce hematoma growth. Sensitivity was estimated. Sensitivity or true positive rate is defined as, the number of strokes correctly identified as spot positive according to the "gold standard" / the total number of strokes identified as spot positive
Time Frame: Baseline head CT scan within 5 hours of stroke, followed by a CT angiogram. Hematoma growth determined by comparison with a head CT scan performed at 24 hours.
Population: The analysis population consists of 19 subjects diagnosed as "Spot Positive" on CT who were eligible for randomization within the clinical trial portion of the protocol, as well as 73 subjects diagnosed as "Spot Negative" on CT who were followed prospectively with no study intervention. Statistical comparison involves only Group 2 and Group 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Randomized to Study Drug | Group 2 - Randomized to Placebo | Group 3 - Observation Only Arm
Number analyzed (Participants) | 10 | 9 | 73
Participants | 4 | 5 | 8
Statistical Analysis 1: Comparison: Group 2 - Randomized to Placebo vs Group 3 - Observation Only Arm; Test type: Superiority; p = 0.004, Fisher Exact; Sensitivity = 38.5, 95% CI 2-sided [17.6 to 64.6]

4. Primary Outcome: The Specificity of the Spot Sign for Predicting Hematoma Growth
Description: The outcome measure is hematoma growth. Groups 2 and 3 only will be compared as group 1 had administration of study drug which was hypothesized to reduce hematoma growth. Specificity was estimated. Specificity or true negative rate is defined as, the number of non-spot positive (spot negative) strokes according to the "gold standard" / the total number of strokes identified as not spot positive.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Randomized to Study Drug | Group 2 - Randomized to Placebo | Group 3 - Observation Only Arm
Number analyzed (Participants) | 10 | 9 | 73
Participants | 4 | 5 | 8
Statistical Analysis 1: Comparison: Group 2 - Randomized to Placebo vs Group 3 - Observation Only Arm; Test type: Superiority; p = 0.004, Fisher Exact; Specificity = 94.2, 95% CI 2-sided [85.6 to 98.1]

5. Secondary Outcome: Number of Participants With Other Potentially Study Drug Related Thromboembolic Complications Such as Deep Venous Thrombosis (DVT) and Elevations in Troponin Not Associated With ECG Changes
Description: Evidence of a deep venous thrombosis or an elevation of troponin within 4 days of completion of study drug administration that are not associated with ECG changes that could be related to the study drug
Time Frame: through day 4 after completion of study drug
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Randomized to Study Drug | Group 2 - Randomized to Placebo | Group 3 - Observation Only Arm
Number analyzed (Participants) | 10 | 9 | 73
Participants | 0 | 1 | 4
Statistical Analysis 1: Comparison: Group 1 - Randomized to Study Drug vs Group 2 - Randomized to Placebo; Test type: Superiority; p = 0.47, Fisher Exact

6. Secondary Outcome: Number of Spot Positive Subjects With 90-day Outcome of Modified Rankin Scale Score >= 5
Description: The modified Rankin Scale (0 is best, 5 is worst - non dead, 6 is dead) was used to define a bad outcome; categorized as a score >=5 versus <5. As the aim of the study was to examine the effect of rFIV!!a only the randomized groups, 1 and 2, defined as spot positive by CTA were compared.
Time Frame: 90 days (+/- 7 days) from time of study enrollment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Randomized to Study Drug | Group 2 - Randomized to Placebo | Group 3 - Observation Only Arm
Number analyzed (Participants) | 10 | 9 | 73
Participants | 3 | 1 | 6
Statistical Analysis 1: Comparison: Group 1 - Randomized to Study Drug vs Group 2 - Randomized to Placebo; Test type: Superiority; p = 0.58, Fisher Exact

7. Secondary Outcome: Number of Participants With Agreement Between the Clinical Site Radiologists and the Study Radiologist With Respect to Identification of a Positive Spot Sign or the Absence of Positive Spot Sign on CTA
Description: The CTA was originally interpreted by the site radiologist so that subjects could be identified as having a positive spot sign for eligibility for randomization. The positive spot sign is indicative that there is potential for further hemorrhagic growth and these subjects were thus eligible to be randomized to receive investigational drug or placebo. The CTA scans were subsequently assessed by the study radiologist and compared for agreement.
Time Frame: Baseline head CT scan within 5 hours, followed by a CT angiogram. Hematoma growth determined by comparison with a head CT scan performed at 24 hours.
Population: The analysis population consists of 19 subjects diagnosed as "Spot Positive" on CT who were eligible for randomization within the clinical trial portion of the protocol, as well as 73 subjects diagnosed as "Spot Negative" on CT who were followed prospectively with no study intervention. Overall agreement was assessed but reported by group below.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Randomized to Study Drug | Group 2 - Randomized to Placebo | Group 3 - Observation Only Arm
Number analyzed (Participants) | 10 | 9 | 73
Participants | 10 | 6 | 69
Statistical Analysis 1: Comparison: Group 1 - Randomized to Study Drug vs Group 2 - Randomized to Placebo vs Group 3 - Observation Only Arm; Test type: Other — A Kappa test of overall agreement was used; Kappa = 0.77, 95% CI 2-sided [0.61 to 0.93] — A kappa of >0.75 is considered excellent agreement

8. Secondary Outcome: Percent Change in Total Hemorrhage Volume (Intracerebral Hemorrhage (ICH) Plus Intraventricular Hemorrhage (IVH)).
Description: Percent change in total volume (intracerebral hemorrhage (ICH) plus intraventricular hemorrhage (IVH)) from baseline CT to 24 hour CT. Percent change is expressed as difference between 24 hour total volume and baseline total volume divided by baseline total volume, expressed as a percentage. In order to examine the effect of rFIVIIa, the randomized groups, Group 1 and Group 2 only were statistically compared.
Time Frame: 24 hours (+/- 3 hours) from baseline CT scan
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline to 24 hours
Arm/Group | Group 1 - Randomized to Study Drug | Group 2 - Randomized to Placebo | Group 3 - Observation Only Arm
Number analyzed (Participants) | 10 | 9 | 73
Percent change from baseline to 24 hours | 13.51 [-0.84 to 33.08] | 20.96 [14.07 to 96.57] | 5.12 [0.28 to 16.64]
Statistical Analysis 1: Comparison: Group 1 - Randomized to Study Drug vs Group 2 - Randomized to Placebo; Groups 1 and 2 only the spot positive subjects randomized to interventional drug or placebo; Test type: Superiority; p = 0.25, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Adverse events were collected out to 90 days from stroke onset
Description: Adverse events and serious adverse events were defined as per clinicaltrials.gov
  A case report form (CRF) was used to collect:
  1. Presence, description and type of adverse events; 2. Severity (mild, moderate, severe, life-threatening, death); 3. Serious (yes, no); 4. Expected (yes, no); 5. Date/Time of onset; 6. Outcome (resolved, continuing, death); 7. Date of resolution; 8. Relation to disease; 9. Relationship to study project; 10. Action taken
Arm/Group | Group 1 - Randomized to Study Drug | Group 2 - Randomized to Placebo | Group 3 - Observation Only Arm
All-Cause Mortality (participants affected / at risk) | 2/10 | 0/9 | 4/73
Serious Adverse Events (participants affected / at risk) | 4/10 | 4/9 | 16/73
Other Adverse Events (participants affected / at risk) | 9/10 | 8/9 | 65/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Randomized to Study Drug (N=10) | Group 2 - Randomized to Placebo (N=9) | Group 3 - Observation Only Arm (N=73)
Cerebral Edema (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
New onset Afib (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atreriovenous malformation (AVM) (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 3 (3) — One not seen on baseline imaging, one complex
Oropharyngeal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ventilator aquired pneuminia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gram negative bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY DISTRESS SECONDARY TO TRACH OBSTRUCTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Elevated Troponin (Investigations) | 1 (1) | 0 (0) | 0 (0)
Left acute on chronic subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — the term was taken directly from the adverse event CRF
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Weakness left leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) — Includes "seizure activity" in Group 1 and "possible simple partial seizure" in Group 3
Slurred speech (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Increasing mass effect (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
POSSIBLE MCA VESSEL THROMBOSIS WITHOUT ISCHEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Significant expansion of ICH (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) — includes "EXACERBATION OF INTRACEREBRAL HEMORRHAGE" in Group 1
Cortical vein thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurologic deterioration (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Neuroleptic malignant syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
WORSENING PERIHEMATOMAL EDEMA AND INCREASING MIDLINE SHIFT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Acute exacerbation of renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
O2 desats on ventilator (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) — Includes "DEPRESSED MENTAL STATUS SECONDARY TO ICH/IVH"
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (DVT) (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) — including one "right iliofemoral DVT"
Hemorrhage expansion (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
PE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Randomized to Study Drug (N=10) | Group 2 - Randomized to Placebo (N=9) | Group 3 - Observation Only Arm (N=73)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) — Mild in group 1
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (6) | 2 (2) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4)
Distended abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 14 (14)
Rectal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) — Group 1 due to hemorrhoids
Chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Fever (General disorders) | 3 (3) | 3 (4) | 6 (6)
Generalized pain (General disorders) | 1 (1) | 1 (1) | 7 (7)
Pain with catherization (General disorders) | 1 (1) | 0 (0) | 0 (0)
Right hand PIV infultration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) — Group1 - oral
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 1 (1) | 12 (13)
Bruising on forearms (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) — Group 1- on forearms Group 3 - on thigh
Fall from bed (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
ELEVATED ERYTHROCYTE SEDIMENTATION RATE (Investigations) | 1 (1) | 0 (0) | 0 (0)
Elevated troponin (Investigations) | 1 (1) | 2 (2) | 5 (5)
Prolonged prothrombin time (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 13 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 17 (17)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 4 (4)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2) — Group 1 right leg Group 2 right knee Group 3 "right knee arthralgia/effusion"
Right shoulder rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aneurysm (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) — Group 1 "SMALL SACCULAR ANEURYSM BASILAR ARTERY" and "ANEURYSM LEFT INTERNAL CAROID ARTERY" same subject
Headache (Nervous system disorders) | 5 (6) | 4 (4) | 11 (11)
Somulence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) — Group1 - increasing Group 2 - persistence
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 5 (5)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Group1 - exacerbation in one subject
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retension (Renal and urinary disorders) | 3 (3) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 1 (1) — Group1 - "PLEURAL EFFUSION, ATELECTASIS" Group 2 "SMALL BILATERAL PLEURAL EFFUSIONS"
Hypertension (Vascular disorders) | 5 (5) | 4 (4) | 32 (32)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
SIADH (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Shivering (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ventriculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
T wave inversion (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3)
hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Asymptomatic MRI DWI lesion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral edema / hydrocephalus (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Confused speech (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Difficult to arouse (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3) — Group 3 - one subject "seizure post (after) arteriovenous malformation repair" Group 3 - one subject "SIMPLE PARTIAL SEIZURES" and "EXACERBATION OF SIMPLE PARTIAL SEIZURE"
Agitation (Psychiatric disorders) | 0 (0) | 2 (2) | 7 (8)
Alcohol withdrawal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) — Group 2 - intermittent
Altered mental status (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) — Group 2 -worsening
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin breakdown / irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 7 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No